CLINICAL TRIAL: NCT01021267
Title: Clinical Pilot Trial on the Influence of a Saw Palmetto Berry Preparation on Sexual Functions in Patients With Benign Prostatic Hyperplasia
Brief Title: Clinical Study to Assess the Influence of a Saw Palmetto Preparation in Patients With Benign Prostatic Hyperplasia (BPH) and Sexual Dysfunctions
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: A. Vogel AG (Industry)
Collaborators: University of London (Other)
Responsible Party: Andy Suter, Head of Med. Dept., Bioforce AG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 920136
Record Dates: First submitted 2009-11-25; First posted 2009-11-26 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Sexual Dysfunctions in Men With Benign Prostatic Hyperplasia
Keywords: sexual dysfunctions; benign prostatic hyperplasia; saw palmetto
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — saw palmetto extract; Prostasan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Saw palmetto berry extract (Experimental): Saw palmetto berry extract, organic saw palmetto, ethanolic extract 96%
  Interventions: Drug: Saw palmetto berry extract

INTERVENTIONS:
Drug: Saw palmetto berry extract — 1x daily 1 capsule containing 320mg lipophilic extract
  Other Names: Prostasan

SUMMARY:
Assessment in an open trial if a standardized saw palmetto preparation has a positive influence on sexual dysfunctions in patients with BPH and sexual dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BPH and sexual dysfunctions (erectile dysfunction or decrease in libido)
* IPSS > 4
* BSFI, sexual drive questions < 5

Exclusion Criteria:

* Lack of libido which is due to a psychic disease or a depressive mood -Excessivly strong lack of libido in the judgement of the investigator within the last two months
* Patients with severe vascular disorders (microangiopathies)
* Patients with known neuropathies
* Severe diabetes mellitus
* Patients with hypertension who are for less than two months on a stable antihypertensive medication
* Known bad compliance of the patient

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Change of the brief Sexual Function Inventory | day 0 and day 56

SECONDARY OUTCOMES:
change in IPSS change in Urolife Quality of Life questionnaire | day 0 and day 56

CONTACTS AND LOCATIONS:
Overall Officials: Eugen Riedi, MD, Principal Investigator — independent
Locations (1):
- Dr. Eugen Riedi, Chur, Switzerland